CLINICAL TRIAL: NCT02353169
Title: The Effects of Dexmedetomidine on Myocardial Repolarization in Children
Brief Title: The Effects of Dexmedetomidine on the Heart Beat During Elective Surgery in Children
Acronym: DexmedQT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Simon Whyte, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: H14-03274
Record Dates: First submitted 2014-12-23; First posted 2015-02-02 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Myocardial Repolarization; Healthy
Keywords: changes in myocardial repolarization in healthy children
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dexmedetomidine 0.25mcg/kg (Experimental): 0.25mcg/kg dexmedetomidine diluted with normal saline in a 10mL syringe, administered intravenously over 60 seconds starting 3 minutes after induction of anesthesia.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.5mcg/kg (Experimental): 0.5mcg/kg dexmedetomidine diluted with normal saline in a 10mL syringe, administered intravenously over 60 seconds starting 3 minutes after induction of anesthesia.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine 0.75mcg/kg (Experimental): 0.75mcg/kg dexmedetomidine diluted with normal saline in a 10mL syringe, administered intravenously over 60 seconds starting 3 minutes after induction of anesthesia.
  Interventions: Drug: Dexmedetomidine
- Saline bolus (Sham Comparator): 10mL normal saline solution administered intravenously over 60 seconds starting 3 minutes after induction of anesthesia.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Precedex
  Arms: Dexmedetomidine 0.25mcg/kg; Dexmedetomidine 0.5mcg/kg; Dexmedetomidine 0.75mcg/kg
Drug: Saline
  Other Names: 9% NaCl
  Arms: Saline bolus

SUMMARY:
Dexmedetomidine is a sedative drug that is commonly used to improve calmness and reduce pain in children waking up after surgery. Some of the side effects of dexmedetomidine, such as a potential change in how the heart muscles contract and changes in blood sugar and potassium levels, are poorly understood. The current study aims to examine these changes directly in healthy children undergoing elective surgery by measuring the heart beats (with an electrocardiogram) and blood sugar and potassium at specific times before and after dexmedetomidine is given. The investigators aim to establish a better understanding of this drug's safety profile.

DETAILED DESCRIPTION:
Purpose:

This study is being conducted to evaluate the effect of three different doses of dexmedetomidine (Precedex® , Hospira Healthcare) on myocardial repolarization, and blood glucose and potassium levels in children undergoing elective surgery.

Hypotheses:

The investigators hypothesize that administering a dexmedetomidine bolus will have some effect on myocardial repolarization, blood glucose, and potassium concentrations in a dose-dependent manner, whereas a saline bolus will not.

Justification:

Dexmedetomidine is a potent, centrally acting α-2 adrenoreceptor agonist with sympatholytic, sedative, amnestic, anxiolytic and analgesic effects, which properties make it popular for use in both pediatric anesthesia and intensive care. In 2013, dexmedetomidine was added to the "possible risk factor for torsades de pointes (TdP)" drug list on crediblemeds.org. Clinicians are currently advised to be vigilant about potential QT prolongation with dexmedetomidine, especially in patients with congenital long QT syndrome (LQTS). However, current evidence for dexmedetomidine-induced prolonged QT is sparse and somewhat contradictory, and the effect of dexmedetomidine on the Tp-e interval has yet to be reported in detail in adults or children. Another poorly defined pharmacodynamic effect of dexmedetomidine is its effect on blood glucose concentration. Theoretically, dexmedetomidine would be expected to cause hypoinsulinaemia and a resultant increase in blood glucose levels (hyperglycemia). Previous studies are in contrast to this however; with reports of hypoglycemia after large doses of the drug. Considering the use of dexmedetomidine in pediatric anesthesia, pediatric intensive care and its increasing use in the neonatal population, increased knowledge of the effect of dexmedetomidine on blood glucose would be valuable.

Finally, hypokalemia is listed as a treatment-emergent adverse event occurring in >2% of adult patients receiving dexmedetomidine in long-term intensive care unit sedation studies. The effect of dexmedetomidine on serum potassium levels in healthy children has yet to be elucidated. Given that hypokalemia increases the risk of TdP, and that there is a possibility that dexmedetomidine may be torsadogenic, this effect is also worthy of investigation.

In sum, the use of dexmedetomidine is associated with many clinical benefits, but its effects on indices of myocardial repolarization, as well as its effects on glucose and potassium metabolism, remain poorly understood and need to be better defined in order to use this drug safely and effectively.

Objectives:

The primary objective of this study is to investigate the effects of three different doses of dexmedetomidine (0.25/0.5/0.75 mcg/kg) on indices of myocardial repolarization (QTc and Tp-e intervals). As a secondary objective, this study will also sample blood glucose and potassium levels before and after dexmedetomidine administration to ascertain if there is any significant effect of a single bolus dose on blood glucose concentrations.

Research Method:

The investigators propose a randomized, single-blinded, 4-group comparative study to characterize the effects of different doses of dexmedetomidine on myocardial repolarization and blood glucose levels in healthy children undergoing elective surgery. The study-specific interventions will include giving a bolus of dexmedetomidine (0.25/0.5/0.75 mcg/kg; or 10mL saline) after induction of general anesthesia, recording two 12-lead ECGs (one before and one after dexmedetomidine administration), and taking three venous blood samples (one before and two after dexmedetomidine administration) to measure glucose and potassium. If the anesthetist would like to administer dexmedetomidine to a participant in the control (saline) group as part of their normal practice, they can do so after the study period is over (after the last blood sample).

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status I-II
* Age 3 to 10yrs
* Elective surgical procedure requiring general anesthesia
* Use of dexmedetomidine acceptable to the staff anesthesiologist
* Un-premedicated
* Ability to read and understand English (parent/legal guardian(s) and child)

Exclusion Criteria:

* Long QT syndrome (LQTS)
* Cardiac disease or rhythm abnormalities
* Family history of LQTS or abnormal cardiac conduction
* Currently taking medications known to prolong QT
* Currently taking medications known to predispose to hypokalemia
* Known hypersensitivity to dexmedetomidine or other study medication
* Weight < 5th centile or > 95th centile for age
* Previously diagnosed hypokalemia
* Impaired renal or liver function
* Pre-operative anxiety requiring sedatives or opioids
* Refusal to participate

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2015-09; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Whyte, MBBS, FRCA, Principal Investigator — BC Children's Hospital, Department of Anesthesia
Locations (1):
- BC Children's Hospital - Department of Anesthesia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorges M, Poznikoff AK, West NC, Brodie SM, Brant RF, Whyte SD. Effects of Dexmedetomidine on Blood Glucose and Serum Potassium Levels in Children Undergoing General Anesthesia: A Secondary Analysis of Safety Endpoints During a Randomized Controlled Trial. Anesth Analg. 2019 Oct;129(4):1093-1099. doi: 10.1213/ANE.0000000000004154. PMID 31008751
- [Derived] Gorges M, Sherwin ED, Poznikoff AK, West NC, Brodie SM, Whyte SD. Effects of Dexmedetomidine on Myocardial Repolarization in Children Undergoing General Anesthesia: A Randomized Controlled Trial. Anesth Analg. 2019 Oct;129(4):1100-1108. doi: 10.1213/ANE.0000000000004135. PMID 30985379

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexmedetomidine 0.25mcg/kg: 0.25mcg/kg dexmedetomidine diluted with normal saline in a 10mL syringe, administered intravenously over 60 seconds starting 3 minutes after induction of anesthesia.
  Dexmedetomidine
- Dexmedetomidine 0.5mcg/kg: 0.5mcg/kg dexmedetomidine diluted with normal saline in a 10mL syringe, administered intravenously over 60 seconds starting 3 minutes after induction of anesthesia.
  Dexmedetomidine
- Dexmedetomidine 0.75mcg/kg: 0.75mcg/kg dexmedetomidine diluted with normal saline in a 10mL syringe, administered intravenously over 60 seconds starting 3 minutes after induction of anesthesia.
  Dexmedetomidine
- Saline Bolus: 10mL normal saline solution administered intravenously over 60 seconds starting 3 minutes after induction of anesthesia.
  normal saline solution
Period: Overall Study
Arm/Group | Dexmedetomidine 0.25mcg/kg | Dexmedetomidine 0.5mcg/kg | Dexmedetomidine 0.75mcg/kg | Saline Bolus
Started | 15 | 18 | 16 | 15
Completed | 12 | 12 | 12 | 12
Not Completed | 3 | 6 | 4 | 3
Not completed — QTc > 450 msec | 1 | 1 | 1 | 1
Not completed — OR team declined | 2 | 0 | 0 | 0
Not completed — Inhalational induction | 0 | 2 | 0 | 0
Not completed — ECG data error | 0 | 3 | 2 | 2
Not completed — Pre-op medication | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine 0.25mcg/kg | Dexmedetomidine 0.5mcg/kg | Dexmedetomidine 0.75mcg/kg | Saline Bolus | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 12 | 12 | 48
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 4.5 [3 to 6.2] | 4.5 [3.8 to 6.5] | 5 [3.8 to 6] | 4.5 [3 to 6] | 5 [3 to 6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 6 | 19
  Male | 9 | 7 | 7 | 6 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 12 | 12 | 12 | 48
Heart Rate (beats/min) [Mean (Standard Deviation); unit: beats/min] | 88.9 (17.8) | 85.7 (13.4) | 84.6 (12.2) | 80.7 (12.5) | 85.0 (14.0)
Corrected QT interval (ms) [Mean (Standard Deviation); unit: ms] | 404.9 (17.1) | 408.8 (15.2) | 409.5 (17.2) | 404.0 (24.1) | 406.8 (18.2)
Interval between the peak and the end of the ECG T wave (Tp-e) [Mean (Standard Deviation); unit: ms] | 66.7 (7.2) | 63.0 (9.4) | 62.8 (6.1) | 65.3 (5.2) | 64.4 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Repolarization (QTc and TP-e Intervals) 1min After Intervention
Description: Absolute QTc and TP-e values 1min after a bolus of dexmedetomidine or saline. Measured with 12-lead ECG.
Time Frame: 60 seconds post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Dexmedetomidine 0.25mcg/kg | Dexmedetomidine 0.5mcg/kg | Dexmedetomidine 0.75mcg/kg | Saline Bolus
Number analyzed (Participants) | 12 | 12 | 12 | 12
ms
  Tp-e Post-intervention | 67.8 (6.0) | 64.0 (10.0) | 64.3 (6.9) | 66.3 (5.9)
  QTc Post-intervention | 395.9 (16.1) | 390.2 (24.0) | 395.4 (18.7) | 416.4 (23.3)

2. Secondary Outcome: Blood Glucose Levels at 15min and 30min Post-intervention
Description: Blood glucose levels at 15 min and 30 min after a bolus of dexmedetomidine or saline. Measured from 1 mL venous blood sample with blood gas analyzer.
Time Frame: over 30 minutes post-intervention
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dexmedetomidine 0.25mcg/kg | Dexmedetomidine 0.5mcg/kg | Dexmedetomidine 0.75mcg/kg | Saline Bolus
Number analyzed (Participants) | 12 | 12 | 12 | 12
mmol/L
  Glucose 15 minutes after intervention | 5.3 (0.7) | 5.6 (0.7) | 5.9 (0.7) | 4.9 (0.7)
  Glucose 30 minutes after intervention | 5.0 (0.7) | 5.0 (0.7) | 5.5 (0.6) | 5.1 (0.7)

3. Secondary Outcome: Blood Potassium Levels at 15min and 30min Post-intervention
Description: Blood potassium levels at 15 min and 30 min after a bolus of dexmedetomidine or saline. Measured from 1mL venous blood sample with blood gas analyzer
Time Frame: over 30 minutes post-intervention
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Dexmedetomidine 0.25mcg/kg | Dexmedetomidine 0.5mcg/kg | Dexmedetomidine 0.75mcg/kg | Saline Bolus
Number analyzed (Participants) | 12 | 12 | 12 | 12
mEq/L
  Potassium 15 minutes after intervention | 3.8 (0.7) | 3.7 (0.2) | 3.8 (0.2) | 3.9 (0.4)
  Potassium 30 minutes after intervention | 3.6 (0.3) | 3.6 (0.4) | 3.8 (0.2) | 3.8 (0.2)

ADVERSE EVENTS:
Time Frame: 30 minutes post-intervention
Description: Serious adverse drug reactions were defined as: hypo-/hypertension requiring intervention; bradycardia, atrioventricular block, or sinus arrest requiring cardiopulmonary resuscitation; or anaphylactic reaction requiring intervention.
Arm/Group | Dexmedetomidine 0.25mcg/kg | Dexmedetomidine 0.5mcg/kg | Dexmedetomidine 0.75mcg/kg | Saline Bolus
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/18 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/18 | 0/16 | 0/15

LIMITATIONS AND CAVEATS:
Healthy children were examined in this study, thus our findings should not be extrapolated to children with long QT syndrome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT02353169/Prot_SAP_000.pdf